CLINICAL TRIAL: NCT07324941
Title: The Role of Electroencephalography Evaluation in Caffeine Discontinuation Timing in Premature Infants
Brief Title: The Role of Electroencephalography in Caffeine Discontinuation Timing in Premature Infants
Status: Not yet recruiting | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Salih Çağrı Çakır, Associate professor, Uludag University
Other Study IDs: 2025/902/17-23
Record Dates: First submitted 2025-12-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Apnea Neonatal; Apnea of Prematurity
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to investigate whether functional maturation assessment by electroencephalography in preterm infants can provide reliable data for the safe discontinuation of caffeine therapy without recurrence of apnea.

In preterm infants receiving caffeine therapy, an assessment of maturation will be performed by EEG at the time when discontinuation of caffeine treatment is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born before 28 weeks of gestation with a birth weight of 1250 grams or less, who received prophylactic caffeine therapy.
2. Infants with a birth weight greater than 1250 grams and a gestational age below 32 weeks, who required invasive mechanical ventilation and were started on prophylactic caffeine therapy.
3. Infants born at less than 37 weeks of gestation, admitted to the neonatal intensive care unit, and treated with caffeine for apnea of prematurity.
4. Infants whose parents or legal guardians provided informed consent.

Exclusion Criteria:

1. Infants who did not receive caffeine therapy,
2. Infants for whom an EEG could not be performed,
3. Infants with major congenital malformations such as neuromuscular disorders, central nervous system developmental abnormalities, thoracic malformations, or major cardiac anomalies,
4. Infants who were transferred to another facility within one week before or after discontinuation of caffeine therapy.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants admitted to the neonatal intensive care unit, born at less than 37 weeks of gestation and receiving caffeine therapy, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of apnea risk after discontinuation of caffeine therapy in preterm infants. | From enrollment to the end of treatment at 4 weeks
  Apnea of prematurity is defined as a sudden cessation of breathing lasting at least 20 seconds, or of shorter duration if accompanied by bradycardia, cyanosis, pallor, or marked hypotonia.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neonatology, Department of Pediatrics, Bursa Uludağ University Faculty of Medicine, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I am not authorized to share patient data.

REFERENCES:
- [Background] Urru SA, Geist M, Carlinger R, Bodrero E, Bruschettini M. Strategies for cessation of caffeine administration in preterm infants. Cochrane Database Syst Rev. 2024 Jul 24;7(7):CD015802. doi: 10.1002/14651858.CD015802.pub2. PMID 39045901
- [Background] Dodson A, Campbell F. Biotin inclusions: a potential pitfall in immunohistochemistry avoided. Histopathology. 1999 Feb;34(2):178-9. No abstract available. PMID 10064400
- [Background] Nayak CS, Anilkumar AC. Neonatal EEG. 2024 Feb 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536953/ PMID 30725638
- [Background] Stevenson NJ, Oberdorfer L, Koolen N, O'Toole JM, Werther T, Klebermass-Schrehof K, Vanhatalo S. Functional maturation in preterm infants measured by serial recording of cortical activity. Sci Rep. 2017 Oct 11;7(1):12969. doi: 10.1038/s41598-017-13537-3. PMID 29021546
- [Background] Shah NA, Wusthoff CJ. How to use: amplitude-integrated EEG (aEEG). Arch Dis Child Educ Pract Ed. 2015 Apr;100(2):75-81. doi: 10.1136/archdischild-2013-305676. Epub 2014 Jul 17. PMID 25035312
- [Background] Gettings JV, Soul JS. Updates in Neonatal Seizures. Clin Perinatol. 2025 Jun;52(2):375-393. doi: 10.1016/j.clp.2025.02.008. Epub 2025 Apr 1. PMID 40350217
- [Background] McCoy B, Hahn CD. Continuous EEG monitoring in the neonatal intensive care unit. J Clin Neurophysiol. 2013 Apr;30(2):106-14. doi: 10.1097/WNP.0b013e3182872919. PMID 23545760
- [Background] Shany E, Berger I. Neonatal electroencephalography: review of a practical approach. J Child Neurol. 2011 Mar;26(3):341-55. doi: 10.1177/0883073810384866. PMID 21383227
- [Background] Koolen N, Dereymaeker A, Rasanen O, Jansen K, Vervisch J, Matic V, De Vos M, Naulaers G, Van Huffel S, Vanhatalo S. Data-driven metric representing the maturation of preterm EEG. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:1492-5. doi: 10.1109/EMBC.2015.7318653. PMID 26736553
- [Background] Bourel-Ponchel E, Gueden S, Hasaerts D, Heberle C, Malfilatre G, Mony L, Vignolo-Diard P, Lamblin MD. Normal EEG during the neonatal period: maturational aspects from premature to full-term newborns. Neurophysiol Clin. 2021 Jan;51(1):61-88. doi: 10.1016/j.neucli.2020.10.004. Epub 2020 Nov 22. PMID 33239230
- [Background] Kaminska A, Eisermann M, Plouin P. Child EEG (and maturation). Handb Clin Neurol. 2019;160:125-142. doi: 10.1016/B978-0-444-64032-1.00008-4. PMID 31277843
- [Background] Muller-Putz GR. Electroencephalography. Handb Clin Neurol. 2020;168:249-262. doi: 10.1016/B978-0-444-63934-9.00018-4. PMID 32164856
- [Background] Jost K, Datta AN, Frey UP, Suki B, Schulzke SM. Heart rate fluctuation after birth predicts subsequent cardiorespiratory stability in preterm infants. Pediatr Res. 2019 Sep;86(3):348-354. doi: 10.1038/s41390-019-0424-6. Epub 2019 May 13. PMID 31086292
- [Background] Jiang JK, Wang C. Maturational delay in the brainstem auditory pathway of very preterm babies with apnoea. Early Hum Dev. 2025 Jan;200:106164. doi: 10.1016/j.earlhumdev.2024.106164. Epub 2024 Nov 28. PMID 39616826
- [Background] Ozkan H, Erdeve O, Kutman HGK. Turkish Neonatal Society guideline on the management of respiratory distress syndrome and surfactant treatment. Turk Pediatri Ars. 2018 Dec 25;53(Suppl 1):S45-S54. doi: 10.5152/TurkPediatriArs.2018.01806. eCollection 2018. PMID 31236018
- [Background] Kaempfen S, Hug M, Sanchez C, Delgado-Eckert E, Schulzke SM. Heart Rate Variability Does Not Predict Recurrence of Apnoea of Prematurity After Ceasing Caffeine Therapy: A Prospective Cohort Study. Acta Paediatr. 2025 Jun;114(6):1371-1378. doi: 10.1111/apa.17579. Epub 2025 Jan 13. PMID 39805735
- [Background] Thompson L, Werthammer JW, Gozal D. Apnea of Prematurity and Oxidative Stress: Potential Implications. Antioxidants (Basel). 2024 Oct 27;13(11):1304. doi: 10.3390/antiox13111304. PMID 39594446
- [Background] Ji D, Smith PB, Clark RH, Zimmerman KO, Laughon M, Ku L, Greenberg RG. Wide variation in caffeine discontinuation timing in premature infants. J Perinatol. 2020 Feb;40(2):288-293. doi: 10.1038/s41372-019-0561-0. Epub 2019 Nov 22. PMID 31758062
- [Background] Acunas B, Uslu S, Bas AY. Turkish Neonatal Society guideline for the follow-up of high-risk newborn infants. Turk Pediatri Ars. 2018 Dec 25;53(Suppl 1):S180-S195. doi: 10.5152/TurkPediatriArs.2018.01817. eCollection 2018. PMID 31236031